CLINICAL TRIAL: NCT03676816
Title: Vaginal Self-sampling for Rapid Turnaround Gonorrhea/Chlamydia Testing in the Emergency Department
Brief Title: Self Sampling for Rapid Turnaround Testing in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Central California Faculty Medical Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018045
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Chlamydia Trachomatis; Neisseria Gonorrhoeae
Keywords: Chlamydia; Gonorrhea
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaginal self-sampling and provider performed endocervical sampling (Experimental): Patients will take part in both provider-performed endocervical sampling (standard care) and vaginal self-sampling.
  Interventions: Procedure: vaginal self sampling; Procedure: provider-performed endocervical sampling

INTERVENTIONS:
Procedure: vaginal self sampling — This is a prospective, non-inferiority trial comparing two methods of collection using a US Food and Drug Administration- cleared 90-minute rapid nucleic acid amplification assay, the Xpert CT/NG assay. Any adult female patient admitted to the Emergency Department at Community Regional Medical Center felt by the provider to require gonorrhea/chlamydia endocervical testing may be entered in the study.
  Other Names: Cepheid, SWAB/A-50
Procedure: provider-performed endocervical sampling — provider-performed endocervical sampling is the gold standard for both gonorrhea and chlamydia. The provider takes a endocervical sample which will get sent to the laboratory as the standard care in comparison to the device being studied.

SUMMARY:
Consenting adult female patient felt by the provider to require gonorrhea/chlamydia endocervical testing will be asked to provide an additional self sample specimen. The specimen will be sent to the laboratory using conventional diagnostic test for gonorrhea/chlamydia.

DETAILED DESCRIPTION:
Study protocol:

1. Initial emergency department history and physical examination (standard procedure).

   a. Provider identifies patient who is felt to require gonorrhea/chlamydia testing.

   i. Provider will contact study staff to consent patient. b. Study staff identifies patient who is felt by provider to require gonorrhea/chlamydia testing. i. Study staff will ask provider if they could move forward with consenting patient.

   c. Provider who is study staff identifies patient who is felt to require gonorrhea/chlamydia testing.
2. Study staff will attempt to consent patient.

   1. If inclusion criteria are met, and there are no exclusion criteria, written informed consent is obtained.
   2. If the patient changes her mind and refuses consent at this point, a notation is written on the front of the research packet, and it is turned in with a refusal notice on the packet.

      * If patient refuses to participate in the self-sampling portion of the study, we will ask patients if they would like to fill out the first half of the patient survey that will contain no personal identification information besides their initials.
3. If patient agrees to participate in the self-sampling, the patient is asked to fill out both page one and page two of the survey after consent is obtained.
4. An attempt is made to write down at least two contact telephone numbers for patients who have given informed consent on page 2 of the patient survey.
5. The patient obtains vaginal self-sample in the restroom/exam room.

   1. A preprinted single-use instruction sheet is given to patient detailing sample collection.
   2. Vaginal self-sampling collection container has preprinted instructions/requisition and a preprinted label on the Cepheid sample tube to the lab denoting this as research sample.
   3. Paper requisition form is also included with the sample which helps with documentation and assigning this sample to be billed to the research study and not to the patient.
   4. The patient returns the collection container after obtaining the sample to study staff that consented the patient.
   5. The collection container will be sent to the lab via pneumatic tube station.
   6. Vaginal self-sampling result is documented in Epic with designation showing differentiation from provider-performed endocervical sampling.
6. Provider-performed endocervical sampling is performed once the patient is assigned a provider and given a private area to conduct a provider-performed endocervical sampling (standard procedure).

   a. The collection container is sent to the lab, and the final result is noted in the medical record as per standard practice (standard procedure).
7. Retrospective chart review is performed three days after patient consented in order to obtain provider-performed endocervical sampling results.
8. Patient will be contacted only if there is a false-negative. A positive with either the self-sample or provider collected sample is considered positive, and patient will not be called back about that

ELIGIBILITY:
Inclusion Criteria:

* Adult female emergency department patient felt by the provider to require gonorrhea/chlamydia endocervical testing

Exclusion Criteria:

* Non-English speakers with the exception of Spanish speakers (once a Spanish-language informed consent document is approved by the Community Medical Center Institutional Review Board)
* Prisoner
* Age <18 years old
* Active psychiatric condition felt to preclude the ability to give informed consent
* Treated for gonorrhea/chlamydia within previous four weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Noninferiority of vaginal self-sampling compared to provider performed endocervical sampling for gonorrhea/chlamydia diagnosis | 2-3 days
  In order for vaginal self-sampling to be considered clinically noninferior to the standard provider-performed endocervical sampling method of collection, we established a minimum sensitivity of 90%. This was based on previous research showing Sexually Transmitted Infection (STI) clinicians' top priority for a point of care STI test is a minimum sensitivity of 90%. In addition, a previous ED study examining urine gonorrhea/chlamydia diagnosis using the same point of care test as this study also used a minimum sensitivity of 90%. (9) Thus, our primary outcome measure was examining for the noninferiority of VSS sensitivity for gonorrhea/chlamydia, with noninferiority being demonstrated if the sensitivity is >=90%.

SECONDARY OUTCOMES:
Predictive value | 2-3 days
  Vaginal self-sampling specificity, positive predictive value, negative productive value for gonorrhea/chlamydia (measured by individual patient)
Predictive value-Gonorrhea | 2-3 days
  Vaginal self-sampling sensitivity, specificity, positive predictive value, negative predictive value for gonorrhea
Predictive value-Chlamydia | 2-3 days
  Vaginal self-sampling sensitivity, specificity, positive predictive value, negative predictive value for chlamydia
Demographics | 2-3 days
  Concordance of vaginal self-sampling to provider-performed endocervical sampling
Percentage | 2-3 days
  Acceptance rate vaginal self-sample
Rate-Worried | 2-3 days
  Rate of patients worried about doing vaginal self-sampling and correctly
Rate-Prefer | 2-3 days
  Rate of patients that prefer vaginal self-sample to provider-performed endocervical sampling
Numeric | 2-3 days
  Number of patients that refused vaginal self-sampling
Descriptive | 2-3 days
  Description of reasons for refusal of vaginal self-sampling

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chinnock, MD, Principal Investigator — UCSF - Fresno
Locations (1):
- Community Regional Trauma and Burn Center, Fresno, California, United States

REFERENCES:
- [Background] Levitt MA, Johnson S, Engelstad L, Montana R, Stewart S. Clinical management of chlamydia and gonorrhea infection in a county teaching emergency department--concerns in overtreatment, undertreatment, and follow-up treatment success. J Emerg Med. 2003 Jul;25(1):7-11. doi: 10.1016/s0736-4679(03)00131-8. PMID 12865101
- [Background] Huppert JS, Taylor RG, St Cyr S, Hesse EA, Reed JL. Point-of-care testing improves accuracy of STI care in an emergency department. Sex Transm Infect. 2013 Sep;89(6):489-94. doi: 10.1136/sextrans-2012-050994. Epub 2013 Mar 7. PMID 23471445
- [Background] Holley CE, Van Pham T, Mezzadra HM, Willis GC, Witting MD. Overtreatment of gonorrhea and chlamydial infections in 2 inner-city emergency departments. Am J Emerg Med. 2015 Sep;33(9):1265-8. doi: 10.1016/j.ajem.2015.06.009. Epub 2015 Jun 12. PMID 26119905
- [Background] Terkelsen D, Tolstrup J, Johnsen CH, Lund O, Larsen HK, Worning P, Unemo M, Westh H. Multidrug-resistant Neisseria gonorrhoeae infection with ceftriaxone resistance and intermediate resistance to azithromycin, Denmark, 2017. Euro Surveill. 2017 Oct;22(42):17-00659. doi: 10.2807/1560-7917.ES.2017.22.42.17-00659. PMID 29067905
- [Background] Katz AR, Komeya AY, Kirkcaldy RD, Whelen AC, Soge OO, Papp JR, Kersh EN, Wasserman GM, O'Connor NP, O'Brien PS, Sato DT, Maningas EV, Kunimoto GY, Tomas JE. Cluster of Neisseria gonorrhoeae Isolates With High-level Azithromycin Resistance and Decreased Ceftriaxone Susceptibility, Hawaii, 2016. Clin Infect Dis. 2017 Sep 15;65(6):918-923. doi: 10.1093/cid/cix485. PMID 28549097
- [Background] Nelson EJ, Maynard BR, Loux T, Fatla J, Gordon R, Arnold LD. The acceptability of self-sampled screening for HPV DNA: a systematic review and meta-analysis. Sex Transm Infect. 2017 Feb;93(1):56-61. doi: 10.1136/sextrans-2016-052609. Epub 2016 Oct 19. PMID 28100761